CLINICAL TRIAL: NCT05893121
Title: Evaluating the Contribution of a Cardiac Coherence Session to Reducing Patients' Anxiety During a Medical Magnetic Resonance Imaging Examination
Brief Title: Evaluation of a Cardiac Coherence Session to Reducing Patients' Anxiety During a MRI Examination
Acronym: RESP-IRM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0483
Record Dates: First submitted 2023-03-20; First posted 2023-06-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
Keywords: cardiac coherence; improving patient management
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: subjects who received information about MRI examination
  Interventions: Other: Information note about MRI
- Experimental: Subjects who received information about MRI examination and one cardiac coherence session
  Interventions: Other: Cardiac coherence session; Other: Information note about MRI

INTERVENTIONS:
Other: Cardiac coherence session — A cardiac coherence session consists of an exercise of six breaths per minute during five minutes.
  Groups: Experimental
Other: Information note about MRI — explanatory note about MRI examination

SUMMARY:
The present project aims at conducting a proof of concept study to explore the pertinence of a single session of cardiac coherence, carried out in patients prior to an MRI examination and presenting anxiety in relation to this examination, to reduce their level of anxiety and thus improve the course of the examination.

DETAILED DESCRIPTION:
Although Magnetic Resonance Imaging (MRI) is considered to be biologically safe and painless, the examination is often perceived by patients as difficult to bear, causing a great deal of anxiety due to the various constraints: the upper half of the body, including the head, positioned in a tube with a circumference of approximately 70 cm, relatively long duration, immobilization and even restraint. However, all these conditions are necessary to obtain good quality images, which are essential for the interpretation of the examination for diagnostic purposes by the clinicians.

The anxiety of patients linked to the performance of an MRI examination and its negative effects are documented in the literature. According to some authors, 71% of the professionals surveyed stated that anxiety was a common problem in their MRI centre and 19% stated that it regularly disrupted the examination. It is estimated that 10% of the motion artefacts present on MRI examinations are caused by anxiety-related motor agitation, making image quality difficult to exploit. Thus, every day, many MRI examinations are cancelled, interrupted, or of poor quality due to movement and difficult to interpret. All these examinations must therefore be rescheduled, with delays that can be several months long.

Among these non-drug methods, cardiac coherence seems promising. This method is recent, non-invasive, of short duration, very easy to implement and requires little training for users.

The present study hypothesize that a single session of cardiac coherence, carried out in patients prior to an MRI examination and presenting anxiety in relation to this examination, could make it possible to reduce their level of anxiety and thus improve the course of the examination.

ELIGIBILITY:
Inclusion Criteria:

* Person affiliated to or benefiting from a social security scheme;
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research);
* Patient to undergo an MRI examination of the upper half of the body
* Patient over 18 years old
* Patient with a high level of anxiety (score ≥ 4) in relation to MRI

Non-inclusion Criteria:

* Patient under legal protection or under another protection regime (guardianship, curatorship).
* Sedated or unconscious patient
* Patient performing an emergency MRI examination
* Patient with a level of French language that does not allow sufficient understanding for the completion of questionnaires

Exclusion criteria:

- STAI Y-A score < 46 (insignificant or low anxiety)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subject with moderate or high anxiety ( score ≥ 4 ) in relation to MRI exam
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Effect of a cardiac coherence session on the anxiety level | 10 minutes
  The anxiety level will be measured by the Y-A form of the Spielberger State-Trait Anxiety Inventory (French version adapted from the "State-Trait Anxiety Inventory" - STAI) in all patients before the MRI examination is performed

SECONDARY OUTCOMES:
MRI examination quality | 30 minutes
  The quality of the MRI examination will be measured at the end of the examination, blinded to the allocation group
Physiological parameters | 30 minutes
  Physiological parameters reflecting the patients' level of anxiety will be measured in all patients before the MRI examination is carried out; before and after reading an information document and performing cardiac coherence for patients in the experimental group, after reading the information document for the control group.
patient satisfaction | 30 minutes
  A satisfaction questionnaire will be used at the end of the MRI examination (2 questions).
Economic evaluation | 30 minutes
  The time spent preparing the patient and the time related to the cardiac coherence consultation
Other economic evaluation | 30 minutes
  The costs related to the imaging act from the point of view of the health insurance

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre DESIRAT, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Pierre Paul Riquet Hospital, Toulouse, France